CLINICAL TRIAL: NCT04434248
Title: An Adaptive, Multicenter, Randomized, Open-label, Comparative Clinical Study to Assess Efficacy and Safety of Favipiravir in Hospitalized Patients With COVID-19
Brief Title: An Adaptive Study of Favipiravir Compared to Standard of Care in Hospitalized Patients With COVID-19
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chromis LLC (Industry)
Collaborators: Chemical Diversity Research Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: COVID-FPR-01
Record Dates: First submitted 2020-06-13; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; 2019-nCoV
MeSH Terms: conditions — COVID-19 | interventions — favipiravir; Standard of Care; Hydroxychloroquine; Chloroquine; Lopinavir; Ritonavir

STUDY DESIGN:
Intervention Model Description: This is an adaptive, multicenter, open-label, randomized clinical study of Favipiravir versus standard of care (SOC) in hospitalized patients with moderate to severe COVID-19 pneumonia.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Favipiravir, lower dose (pilot stage) (Experimental): 1600mg BID on the 1st day followed by 600mg BID for 13 days
  Interventions: Drug: Favipiravir
- Favipiravir, higher dose (pilot stage) (Experimental): 1800mg BID on the 1st day followed by 800mg BID for 13 days
  Interventions: Drug: Favipiravir
- Standard of care (pilot stage) (Active Comparator): Based on approved clinical recommendations for treatment of COVID-19 in the Russian Federation (but not Favipiravir). Might include hydroxychloroquine, chloroquine, lopinavir/ritonavir or other recommended schemes.
  Interventions: Drug: Standard of Care
- Favipiravir, selected dose (pivotal stage) (Experimental): The dose will be selected based on pilot study results.
  Interventions: Drug: Favipiravir
- Standard of care (pivotal stage) (Active Comparator): Based on approved clinical recommendations for treatment of COVID-19 in the Russian Federation (but not Favipiravir). Might include hydroxychloroquine, chloroquine, lopinavir/ritonavir or other recommended schemes.
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: Favipiravir — 200 mg coated tablets
  Other Names: Avifavir
  Arms: Favipiravir, higher dose (pilot stage); Favipiravir, lower dose (pilot stage); Favipiravir, selected dose (pivotal stage)
Drug: Standard of Care — Standard of Care will be prescribed in accordance with the recommended treatment regimens presented in the Russian guidelines for the prevention, diagnosis and treatment of COVID-19 according to the decision of the Investigator.
  Other Names: Hydroxychloroquine, chloroquine, lopinavir/ritonavir, etc.
  Arms: Standard of care (pilot stage); Standard of care (pivotal stage)

SUMMARY:
The study is Phase II/III and consists of pilot and pivotal stages. The objective of the pilot stage is to conduct a preliminary assessment of the efficacy and safety of Favipiravir, and to select the optimal dosing regimen to study during the pivotal stage. The objective of the pivotal stage is to assess the efficacy and safety of Favipiravir compared with the Standard of care (SOC) in hospitalized patients with moderate to severe COVID-19 pneumonia.

DETAILED DESCRIPTION:
At the pilot stage: upon signing the informed consent form and screening, 60 eligible patients with polymerase chain reaction (PCR) confirmed COVID-19 pneumonia are randomized at a 1:1:1 ratio to receive either Favipiravir 1600 mg twice a day (BID) on Day 1 followed by 600 mg BID on Days 2-14 (1600/600 mg), or Favipiravir 1800 mg BID on Day 1 followed by 800 mg BID on Days 2-14 (1800/800 mg), or SOC.

At the pivotal stage: additional 270 eligible patients are randomized at a 1:1 ratio to receive either Favipiravir (the dose regimen depends of the subject's weight) or SOC.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Patient Information Sheet and Informed Consent form to participate in the study.
2. Men and women aged 18 years and older.
3. Patients hospitalized with a diagnosis of COVID-19.
4. The diagnosis of COVID-19 was confirmed by positive reverse transcription polymerase chain reaction (RT-PCR) test for SARS-CoV-2, performed no earlier than 7 days before hospitalization or at screening.
5. Moderate severity of COVID-19 with pneumonia with at least 1 of the following symptoms:

   * Fever above 38 °C;
   * Cough;
   * Shortness of breath during physical exertion;
   * C reactive protein (CRP) of blood serum > 10 mg/l;
   * SpO2 < 95%
6. The capability of oral drug administration.
7. The patients' consent to use adequate contraception methods during the study (condom with spermicide) and for 3 months following completion.

Exclusion Criteria:

1. Severe type of disease, with at least one of the following criteria:

   * Frequency of breath > 35 per minute, which does not decrease after the body temperature drops to normal or subfebrile values;
   * Blood oxygen saturation (SpO2) < 90% at rest;
   * Partial pressure of oxygen in arterial blood (PaO2) < 60 mm Hg;
   * Oxygenation index (RaO2/FiO2) ≤ 200 mm Hg;
   * Partial pressure of CO2 in arterial blood (PaCO2) < 60 mm Hg;
   * Septic shock.
2. Patients treated with lopinavir/ritonavir, ribavirin, arbidol, chloroquine, hydroxychloroquine, mefloquine, favipiravir within 7 days prior to screening.
3. Severe cardiovascular diseases currently or 6 months prior to randomization, including: New York Heart Association (NYHA) Class III or IV chronic heart failure, clinically significant ventricular arrhythmias (ventricular tachycardia, ventricular fibrillation), unstable angina, myocardial infarction, heart and coronary vessel surgery, significant valvular heart disease, uncontrolled arterial hypertension with systolic blood pressure > 180 mm Hg and diastolic blood pressure > 110 mm Hg, pulmonary embolism or deep vein thrombosis.
4. Severe chronic renal impairment (GFR < 30 ml / min) or continuous renal replacement therapy, hemodialysis or peritoneal dialysis.
5. A history of cirrhosis or an increase in alanine aminotransferase (ALT) and / or aspartate aminotransferase (AST) > 5 times × upper limit of normal (ULN).
6. Severe diseases of the central nervous system, including seizures in history or conditions that may lead to their development; stroke or transient ischemic attack within 12 months prior to screening; head injuries or loss of consciousness within 12 months prior to screening; a brain tumor.
7. Significant uncontrolled concomitant disease, e.g. neurological, renal, hepatic, endocrinological or gastrointestinal disorder which according to the Investigator, could prevent the patient from participating in the study
8. Malignancies that require chemotherapy within 6 months prior to screening.
9. Known HIV infection
10. Hypersensitivity to any component of the study drug.
11. Participation in other clinical studies or taking other study drugs within 28 days prior to screening.
12. Pregnant or lactating women or women planning to get pregnant during the clinical study; women of child-bearing potential (including non-sterilized by surgical means and during the post-menopause period less than 2 years) who do not use adequate contraception methods.
13. Inability to read or write, unwillingness to understand and follow procedures of study protocol, as well as any other concomitant medical or serious mental conditions that make the patient unfit to participate in the study, limit the legality of obtaining informed consent or can affect patient's ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Rate of viral elimination by Day 10 [pilot stage, dose selection] | 10 Days
  Percent of patients with undetectable SARS-CoV-2 RNA level on Day 10
Time to viral elimination [pivotal stage] | 28 Days
  Median time to reach undetectable SARS-CoV-2 RNA level
Time to clinical improvement [pivotal stage] | 28 Days
  Median time reach clinical improvement (2 points of the Ordinal Scale for Clinical Improvement) or discharge from the hospital

SECONDARY OUTCOMES:
Rate of viral elimination | Days 3, 5, 7, 9, and 11
  Percent of patients with undetectable SARS-CoV-2 RNA level
Time to normalization of clinical symptoms | 28 Days
  Median time [days] to reach normal levels of clinical indicators (body temperature, SpO2, breathing rate)
Duration of oxygen therapy | 28 Days
  Mean duration of oxygen therapy [days]
Change in the level of lung damage according to CT | Days 15, 22, and 29
  Change of lung damage level according to CT comparing to baseline [% of patients]
Rate of transfer to the intensive care unit | 28 days
  Percent of patients transferred to the intensive care unit [% of patients]
Rate of the use of non-invasive lung ventilation | 28 days
  Percent of patients undergoing non-invasive lung ventilation [% of patients]
Rate of the use of mechanical ventilation | 28 days
  Percent of patients undergoing mechanical ventilation [% of patients]
Mortality | 28 days
  Percent of patients died within 28-days period [% of patients]
Peak plasma concentration (Cmax) | Day 1
  Determination of Cmax [ng/ml]
Time to peak plasma concentration (Tmax) | Day 1
  Determination of Tmax [h]
Area under the plasma concentration versus time curve (AUC0-t) | 10 days
  Determination of AUC0-t [ng*h/ml]
Trough plasma concentration (Ctrough) | 10 days
  Determination of Ctrough [ng/ml]

CONTACTS AND LOCATIONS:
Overall Officials: Elena Pavlikova, MD,PhD,Prof, Principal Investigator — Moscow State University n.a. M.V. Lomonosov; Nikita Lomakin, MD,PhD, Principal Investigator — Central Clinical Hospital with Polyclinic
Locations (22):
- Russia (22):
  - Republican Clinical Hospital, Makhachkala
  - "K+31" Clinic, Moscow
  - "Khaven" Llc, Moscow
  - Central Clinical Hospital with Polyclinic, Moscow
  - Central Research Institute of Epidemiology, Moscow
  - City Clinical Hospital n.a. O.M. Filatov, Moscow
  - City Clinical Hospital named after S.S. Yudin, Moscow
  - City Clinical Hospital No. 24, Moscow
  - City Clinical Hospital No. 51, Moscow
  - First Moscow State Medical University n.a. I.M. Sechenov, Moscow
  - Moscow State University n.a. M. V. Lomonosov, Moscow
  - National Medical and Surgical Center named after N.I. Pirogov, Moscow
  - City Hospital № 33 of the Leninsky region of Nizhny Novgorod, Nizhny Novgorod
  - Infectious clinical hospital No.2 of Nizhny Novgorod, Nizhny Novgorod
  - Ryazan State Medical University named after I.P. Pavlov, Ryazan
  - Military Medical Academy named after S.M. Kirova, Saint Petersburg
  - Saratov State Medical University named after V.I. Razumovsky, Saratov
  - Clinical hospital No.1, Smolensk
  - Regional Clinic Hospital, Tver'
  - Bashkir State Medical University, Ufa
  - Yakutsk City Clinical Hospital, Yakutsk
  - Yaroslavl Regional Clinical Hospital for War Veterans, Yaroslavl

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ivashchenko AA, Dmitriev KA, Vostokova NV, Azarova VN, Blinow AA, Egorova AN, Gordeev IG, Ilin AP, Karapetian RN, Kravchenko DV, Lomakin NV, Merkulova EA, Papazova NA, Pavlikova EP, Savchuk NP, Simakina EN, Sitdekov TA, Smolyarchuk EA, Tikhomolova EG, Yakubova EV, Ivachtchenko AV. AVIFAVIR for Treatment of Patients With Moderate Coronavirus Disease 2019 (COVID-19): Interim Results of a Phase II/III Multicenter Randomized Clinical Trial. Clin Infect Dis. 2021 Aug 2;73(3):531-534. doi: 10.1093/cid/ciaa1176. PMID 32770240